CLINICAL TRIAL: NCT00002688
Title: AML-MVPCYA: ADDITION OF CYCLOSPORIN A TO THE COMBINATION OF MITOXANTRONE AND ETOPOSIDE (VP 16,213) TO OVERCOME RESISTANCE TO CHEMOTHERAPY IN REFRACTORY AML: A RANDOMIZED PHASE II STUDY
Brief Title: Cyclosporine and Combination Chemotherapy in Treating Patients With Relapsed or Refractory Acute Myeloid Leukemia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Medical Center Groningen (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000064413; DUT-KWF-CKVO-9412; EU-95003
Record Dates: First submitted 1999-11-01; First posted 2004-07-29 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2007-05

CONDITIONS: Leukemia
Keywords: recurrent adult acute myeloid leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Acute | interventions — Cyclosporine; Etoposide; Mitoxantrone

INTERVENTIONS:
Drug: cyclosporine
Drug: etoposide
Drug: mitoxantrone hydrochloride

SUMMARY:
RATIONALE: Some cancers become resistant to chemotherapy drugs. Combining cyclosporine with chemotherapy may prevent resistance to the drugs and allow the cancer cells to be killed.

PURPOSE: Randomized phase II trial to study the effectiveness of adding cyclosporine to combination chemotherapy in treating patients with relapsed or refractory acute myeloid leukemia.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate whether the addition of cyclosporine (CYSP) to mitoxantrone (DHAD) and etoposide (VP-16) increases the response rate and duration of response in adults with refractory or relapsed acute myelogenous leukemia (AML). II. Correlate response to this treatment with the presence of P-glycoprotein (P-gp) multidrug resistance (MDR) and the degree of in vitro modulation of leukemic blasts, including CD34+ blasts. III. Correlate response with the presence of other resistance mechanisms, such as atypical MDR and non-P-gp phenotype. IV. Evaluate the toxicity of this treatment in AML patients. V. Study the effect of CYSP on DHAD and VP-16 pharmacokinetics and metabolism and, potentially, on intracellular drug accumulation.

OUTLINE: Randomized study. The following acronyms are used: CYSP Cyclosporine, NSC-290193 DHAD Mitoxantrone, NSC-301739 VP-16 Etoposide, NSC-141540 Arm I: 2-Drug Combination Chemotherapy. DHAD; VP-16. Arm II: 2-Drug Combination Chemotherapy with Drug Resistance Inhibition. DHAD; VP-16; with CYSP.

PROJECTED ACCRUAL: At least 25 patients/arm will be entered over approximately 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Acute myelogenous leukemia (AML) in the following categories: Refractory to initial standard therapy consisting of idarubicin/cytarabine and amsacrin/cytarabine (on protocol HOVON 29) First or subsequent relapse following complete response to standard chemotherapy (on protocols HOVON 4/4A or 11 or any other protocol) At least 6 months between mitoxantrone/etoposide and relapse No myelodysplasia

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Not specified Hematopoietic: Not applicable Hepatic: Bilirubin no greater than 2 x normal Alkaline phosphatase no greater than 2 x normal Renal: Creatinine no greater than 1.7 mg/dl (150 micromoles/liter) OR Creatinine clearance at least 60 ml/min Cardiovascular: No uncontrolled hypertension No other severe cardiac disease Pulmonary: No severe pulmonary disease Other: No known intolerance to any study drug No uncontrolled severe infection Not HIV seropositive No severe neurologic or metabolic disease No concomitant malignancy except: Nonmelanomatous skin cancer In situ cervical carcinoma No pregnant women

PRIOR CONCURRENT THERAPY: See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 1995-02

CONTACTS AND LOCATIONS:
Overall Officials: Simon Daenen, MD, PhD, Study Chair — University Medical Center Groningen
Locations (12):
- Belgium (2):
  - Cliniques Universitaires Saint-Luc, Brussels (Bruxelles)
  - U.Z. Gasthuisberg, Leuven
- Netherlands (7):
  - Leyenburg Ziekenhuis, 's-Gravenhage (Den Haag, the Hague)
  - Academisch Ziekenhuis der Vrije Universiteit, Amsterdam
  - Academisch Medisch Centrum, Amsterdam
  - Academisch Ziekenhuis Groningen, Groningen
  - Academisch Ziekenhuis Maastricht, Maastricht
  - University Hospital - Rotterdam Dijkzigt, Rotterdam
  - Academisch Ziekenhuis Utrecht, Utrecht
- Switzerland (3):
  - University Hospital, Basel
  - Inselspital, Bern, Bern
  - Universitaetsspital, Zurich